CLINICAL TRIAL: NCT03168698
Title: Carbetocin vs. Oxytocin at Elective Cesarean Section: a Double-blind, Randomized Controlled Non-inferiority Trial of High and Low Dose Regimens
Brief Title: Carbetocin vs. Oxytocin at Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-01
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; cesarean delivery; carbetocin; duratocin; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carbetocin 20mcg (Active Comparator): Carbetocin 20mcg, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator): Carbetocin 100mcg, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Carbetocin
- Oxytocin 0.5IU (Active Comparator): Oxytocin 0.5IU, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Oxytocin
- Oxytocin 5IU (Active Comparator): Oxytocin 5IU, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Patient is given carbetocin (20 or 100 mcg) intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Other Names: Duratocin
  Arms: Carbetocin 100mcg; Carbetocin 20mcg
Drug: Oxytocin — Patient is given oxytocin (0.5 or 5 IU) intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Other Names: Pitocin
  Arms: Oxytocin 0.5IU; Oxytocin 5IU

SUMMARY:
The study investigators are comparing 2 drugs (oxytocin and carbetocin) at 2 different dosages, to help prevent serious bleeding (hemorrhage) after cesarean deliveries. These drugs are used routinely to help contract the uterus and keep it contracted after the delivery of the baby and placenta; this reduces the amount of blood you might lose. At Mount Sinai Hospital, currently oxytocin is used, but its effect on the uterus is much shorter than that of carbetocin. Internationally, there is no consensus as to what the most effective drug to use is and at which dose. The Society of Obstetricians and Gynaecologists of Canada has recently revised its guidelines to suggest 100 micrograms (mcg) of carbetocin as the drug of choice at elective cesarean section. Guidelines from the United Kingdom and the United States currently suggest oxytocin at various doses as the drug of choice at elective cesarean sections. Previous studies at Mount Sinai Hospital have shown that lower doses of oxytocin, 0.35 International Units (IU), and carbetocin, 20 mcg, may be as effective as the higher recommended doses. The investigators plan to conduct a large study to confirm these findings so that they can use the most appropriate dose in the future. Furthermore, the investigators hope to demonstrate that side effects are lower with the lower dose regimens.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most commonly used uterotonic drug to prevent and treat PPH in the world. However, oxytocin has a very short duration of action, requiring a continuous infusion to achieve sustained uterotonic activity. Moreover, large doses are associated with adverse effects like hypotension, nausea, vomiting, dysrhythmias and ST changes. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recommended a single dose of 100 mcg of the longer acting carbetocin at elective cesarean section to promote uterine contraction. In multiple studies performed at Mount Sinai Hospital, we have shown that smaller doses of oxytocin (ED 90 0.35 IU) and carbetocin (ED 90 14.8 mcg) are effective in achieving adequate uterine tone at elective cesarean section. No study has directly compared the high dose regimens with the low dose regimens; therefore a large double-blind randomized controlled trial is necessary to show the non-inferiority of the lower doses of both drugs.

There is a lack of consensus as to what the optimal uterotonic regime is globally. Furthermore, variability in the international guidelines regarding the choice of first line uterotonic in prevention of PPH adds to the confusion. With the widespread availability of carbetocin in some of the developed countries, including Canada, the question of which uterotonic to adopt and at which dose becomes even more difficult to ascertain. Studies that have currently been published suggest the ED90 doses of carbetocin and oxytocin provide adequate uterine contraction with possibly fewer side effects associated with the lower dosed regimens. These advantages may provide a better safety profile and patient satisfaction. To the best of our knowledge, no studies have compared the low doses (ED90) of oxytocin vs. carbetocin, or low (ED90) vs high (conventional) doses of the two drugs in the setting of elective cesarean section. The results of this study will provide evidence on the efficacy and safety of the ED90 dosing compared directly to the higher dosing of both drugs.

Our hypothesis is that the ED90 doses of carbetocin and oxytocin will not be inferior to the higher dosing as determined by the intensity of uterine contraction using a VNRS in women undergoing elective cesarean section. We anticipate that the intensity of uterine contraction using the VNRS at 2 minutes post administration of all drugs will fall within the predetermined margin to signify non-inferiority of all regimens.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section under spinal anesthesia.
* Written informed consent to participate in this study.
* Full-term pregnancy
* Non labouring patients

Exclusion Criteria:

* Refusal to give written informed consent.
* Allergy or hypersensitivity to carbetocin or oxytocin.
* Labouring patients
* Need for general anesthesia
* Conditions that predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, preeclampsia, eclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* Hepatic, renal, and cardiovascular disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Uterine Tone 2 minutes | 2 minutes
  Intensity of uterine tone on a VNRS scale of 0-10 as evaluated by the obstetrician at 2 minutes after completion of injection of the bolus study drug.

SECONDARY OUTCOMES:
Uterine Tone 5 minutes | 5 minutes
  Intensity of uterine tone on a VNRS scale of 0-10 as evaluated by the obstetrician at 5 minutes after completion of injection of the bolus study drug.
Uterine Tone 10 minutes | 10 minutes
  Intensity of uterine tone on a VNRS scale of 0-10 as evaluated by the obstetrician at 10 minutes after completion of injection of the bolus study drug.
Additional uterotonics - operating room | 1 hour
  The use of additional uterotonic agents in the operating room
Additional uterotonics - 24 hours | 24 hours
  The use of additional uterotonic agents at any time after admission to the recovery room and up to 24 hours post delivery
Estimated blood loss | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 24 hours after the cesarean section.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Hypertension: systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient
Presence of flushing: questionnaire | 2 hours
  Any presence of flushing, from drug administration until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - McMaster University Medical Centre (MUMC), Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No